CLINICAL TRIAL: NCT06553963
Title: Biochemical Monitoring and Nutritional Support During Pre-Competition Weight Reduction in Female Weightlifters: A Randomized Controlled Trial
Brief Title: Athlete Biochemical Monitoring and Nutritional Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Principal Investigator, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SSC20246
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Weight Reduction
MeSH Terms: conditions — Weight Loss | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): All participants followed their coaches' regular training plans for daily training (actual pre-competition training environment), without altering their personal routines or lifestyle habits.
- Experimental group (Experimental): Participants in the experimental group received a four-week tailored nutrition program, developed by sports nutritionists based on athletes' biochemical profiles, body weight, training intensity, and dietary habits. The program included:
  Daily Dietary Logs: Monitoring food intake for immediate nutritional adjustments.
  Weekly Nutritional Consultations: Strategy refinement discussions with experts. Customized Nutritional Supplements: "Zinc Magnesium Multi-Vitamin Sports Nutrition Powder" was used to improve blood urea, cortisol, and hemoglobin levels, containing ingredients like rice bran lipid alcohol, magnesium, zinc, and B vitamins.
  Performance-Specific Supplements: "Endurance Sugar Pump" to lower creatine kinase levels during training and "Testosterone Synthesis Pump" to enhance testosterone, both by Weite Beijing Co., Ltd.
  Sleep Aid: "Melatonin Tablets" to ensure restful sleep, containing vitamin B6 and melatonin, produced by Dongli Beijing Co., Ltd.
  Interventions: Other: Control group; Other: Experimental group

INTERVENTIONS:
Other: Control group — The control group maintained their regular diet and training without additional nutritional support.
  Arms: Experimental group
Other: Experimental group — Biochemical Monitoring and Nutritional Support
  Arms: Experimental group

SUMMARY:
The objective of this study is to evaluate the efficacy of physiological and biochemical monitoring along with nutritional support in improving the performance and well-being of female weightlifters during the critical weight reduction phase before competition. It also seeks to determine the safety and potential benefits of the personalized nutritional interventions.

The primary questions this study aims to address are:

Does personalized nutritional support, informed by physiological and biochemical monitoring, reduce the incidence of fatigue and improve sleep quality in female weightlifters during the pre-competition period? How do serum indicators change in response to the nutritional interventions, and what does this indicate about the athletes' health and performance? What are the perceived benefits and any potential adverse effects reported by the participants receiving the nutritional support? To assess the impact of the intervention, researchers will compare the outcomes of the experimental group, which receives the tailored nutritional support, to those of the control group, which follows standard practices without additional intervention.

Participants will be required to:

Consume the nutritional supplements or maintain their regular diet as assigned for the duration of the 1-month study.

Attend scheduled visits to the research facility every two weeks for comprehensive health assessments, including blood tests for serum indicators and evaluations of fatigue levels and PSQI scores.

Record their daily experiences, including dietary adherence, training intensity, perceived fatigue, sleep patterns, and any other relevant observations in a personal diary.

By conducting this randomized controlled trial, the study will provide valuable insights into the role of targeted nutritional support in enhancing athletic performance and overall health during the demanding pre-competition weight reduction period.

DETAILED DESCRIPTION:
The study took place from August to September 2024, spanning a total of 4 weeks. Initially, all participants followed their coaches' regular training plans for daily training (actual pre-competition training environment), without altering their personal routines or lifestyle habits.

On this foundation, participants in the experimental group received a four-week personalized nutritional monitoring and supplementation program. This program was tailored by sports nutrition experts according to each athlete's biochemical indicators, body weight, training load, and personal dietary habits. It specifically included, but was not limited to: Nutritional Assessment, where a detailed nutritional evaluation was conducted for each athlete before the start of the study, including dietary history, biochemical indicator analysis, etc.; Dietary Logs, where athletes were asked to record their daily food intake to allow the nutrition team to monitor and adjust in real time; Nutritional Consultations: Weekly face-to-face consultations with nutrition experts to discuss dietary plans and resolve any questions or issues; Nutritional Supplements: Adjusting the types and dosages of nutritional supplements based on weekly biochemical monitoring results, aimed at optimizing athletes' biochemical indicators, such as reducing blood urea and cortisol, and increasing hemoglobin (Nutritional supplement name: Zinc Magnesium Multi-Vitamin Sports Nutrition Powder, 180 g/bag; Origin: Beijing, China, Winpowerdata Technology (Beijing) Co., Ltd.; Ingredients: Rice bran lipid alcohol, magnesium, zinc, vitamin C, taurine, vitamin B1, vitamin B2, vitamin B6; Dosage: 1-2 bags daily); Reducing creatine kinase (Nutritional supplement name: Endurance Sugar Pump, 70 g/bag; Origin: Beijing, China, Weite Beijing Co., Ltd.; Ingredients: Soluble barley starch 62 g, fructose 1,6-diphosphate 6 g, electrolytes; Dosage: 1-2 bags during daily training); Enhancing testosterone (Nutritional supplement name: Testosterone Synthesis Pump, 1 capsule/2 grams; Origin: Beijing, China, Weite Beijing Co., Ltd.; Ingredients: Super testosterone complex, testosterone action amplification factor, testosterone receptor sensitizer, 5-level male testosterone optimization factor, aspartic acid, Rhodiola; Dosage: 6 capsules before daily training); Promoting sleep (Nutritional supplement name: Melatonin Tablets, 1 tablet/0.5 grams; Origin: Beijing, China, Dongli Beijing Co., Ltd.; Ingredients: Vitamin B6, 1600 mg/100 g, melatonin, 500 mg/100 g; Dosage: 1 tablet before bedtime); Control group participants continued to follow their regular diet and training plan without additional nutritional intervention.

This study conducted 5 tests on all participants, at baseline (before weight reduction), week one, week two, week three, and week four (1-2 days before the competition). The time was fixed on Sunday (6:30-7:30 AM). The Pittsburgh Sleep Quality Index (PSQI) test was conducted twice (at baseline and week four).

Serum Testing: Approximately 2 ml of fasting venous blood was taken from the participants' elbow. Beckman Coulter Automated Biochemical Analyzer (California, USA) was used to measure blood urea and creatine kinase, Beckman Coulter Chemiluminescence Immunoassay Analyzer (California, USA) was used to measure blood testosterone and cortisol, and HemoCue Hb 301 Hemoglobinometer (Sweden) was used to measure hemoglobin.

Scale Testing: Participants' fatigue scores were tested, with participants asked to mark their fatigue score on a 10 cm line, with the far left indicating no fatigue and the far right indicating severe fatigue. The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire used to assess the sleep quality of the subject over the past month, composed of 18 self-rated items forming 7 components, with a total score ranging from 0 to 21 points, the higher the score, the worse the sleep quality. The scale's reliability for Chinese subjects is between 0.65 and 0.84, and the validity is greater than 0.85

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years old
* At least 5 years of professional weightlifting training experience
* Currently undergoing systematic training
* Passed a health examination
* The study complies with the Declaration of Helsinki and signed an informed consent form.

Exclusion Criteria:

* Obvious injuries to the lower limb joints
* Taking prescription medications (such as those affecting mood and sleep)
* Abnormal cardiovascular function.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Serum Testing: blood urea | 28 Days
  Approximately 2 ml of fasting venous blood was taken from the participants' elbow. Beckman Coulter Automated Biochemical Analyzer (California, USA) was used to measure blood urea.
Serum Testing: creatine kinase | 28 Days
  Approximately 2 ml of fasting venous blood was taken from the participants' elbow. Beckman Coulter Automated Biochemical Analyzer (California, USA) was used to measure creatine kinase.
Serum Testing: blood testosterone | 28 Days
  Beckman Coulter Chemiluminescence Immunoassay Analyzer (California, USA) was used to measure blood testosterone.
Serum Testing: cortisol | 28 Days
  Beckman Coulter Chemiluminescence Immunoassay Analyzer (California, USA) was used to measure blood cortisol.
Serum Testing: hemoglobin | 28 Days
  HemoCue Hb 301 Hemoglobinometer (Sweden) was used to measure hemoglobin.
Scale Testing: fatigue scores | 28 Days
  Participants were requested to assess their level of fatigue using the Visual Analogue Scale (VAS) for Fatigue, a validated measurement tool. On the VAS, a 10 cm line is marked, where '0' cm represents no fatigue and '10' cm represents the most severe fatigue possible. Higher scores on this scale indicate a greater degree of fatigue, with lower scores reflecting less fatigue.
Scale Testing: Pittsburgh Sleep Quality Index | 28 Days
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire used to assess the sleep quality of the subject over the past month, composed of 18 self-rated items forming 7 components, with a total score ranging from 0 to 21 points, the higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Cheng, Dr, Study Chair — Chengdu Sport University

IPD SHARING:
Plan to Share IPD: No